CLINICAL TRIAL: NCT06724640
Title: A Phase 1 Double-Blind (Sponsor-unblinded), Placebo-Controlled, Randomized, Single Dose Escalation Study to Investigate the Safety, Tolerability, and Pharmacokinetics of Parenterally Administered Long-acting Formulations of VH4011499 in Adults Without HIV
Brief Title: A Study to Assess the Safety, Tolerability, and Pharmacokinetics of VH4011499 Compared to Placebo in Adults Without HIV
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 218547
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: HIV Infections
Keywords: Human Immunodeficiency Virus (HIV); VH4011499; Safety; Tolerability; Pharmacokinetics; Healthy participants; Long-Acting Injection; Single ascending dose; Multiple ascending dose
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single ascending dose (SAD) Group (Experimental): Participants in this group will be randomized to receive a single dose of either VH4011499 low dose or VH4011499 high dose or placebo.
  Interventions: Drug: VH4011499 low dose Injection; Drug: VH4011499 high dose Injection; Drug: Placebo
- Multiple ascending doses (MAD) Group (Experimental): Participants in this group will be randomized to receive two doses of either VH4011499 low dose or VH4011499 high dose or placebo.
  Interventions: Drug: VH4011499 low dose Injection; Drug: VH4011499 high dose Injection; Drug: Placebo

INTERVENTIONS:
Drug: VH4011499 low dose Injection — VH4011499 low dose Injection will be administered subcutaneously and/or intramuscularly.
Drug: VH4011499 high dose Injection — VH4011499 high dose Injection will be administered subcutaneously and/or intramuscularly.
Drug: Placebo — Placebo Injection will be administered either subcutaneously or intramuscularly.

SUMMARY:
The purpose of this study is to investigate safety, pharmacokinetics and tolerability following single ascending dose (SAD) and multiple ascending doses (MAD) of VH4011499 administered subcutaneously (SC) and intramuscularly (IM) in participants without HIV.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 55 years of age inclusive, at the time of signing the informed consent.
* Participants who are overtly healthy.
* Participants may be male or female. Participants assigned female at birth are eligible to participate if they are not pregnant, not planning to become pregnant during the study, not breast/chest feeding or planning to breast/chest feed during the study and one of the following applies:

  * Is a Participant of Nonchildbearing potential (PONCBP)
  * Is a Participant of Childbearing potential (POCBP) and using a highly effective method of contraception through 78 weeks after the last dose of parenteral VH4011499 or through the end of the study. The investigator is responsible for review of medical history, menstrual history and recent sexual activity to decrease the risk for inclusion of a POCBP with an early pregnancy.
* Capable of giving signed informed consent.

Exclusion Criteria:

* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, neurological or psychiatric disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention or interfering with the interpretation of data.
* Abnormal blood pressure.
* Lymphoma, leukemia, or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years.
* Breast cancer within the past 10 years.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities.
* History of clinically relevant hepatitis within last 6 months.
* Patients with chronic hepatitis B infection.
* History of sensitivity to any of the study interventions, a history of drug allergy or other allergy that contraindicates their participation.
* The participant has an underlying skin disease or disorder that would interfere with assessment of injection sites.
* Participants considered to have insufficient musculature to allow safe VH4011499 intramuscular administration will be excluded.
* History of or on-going high-risk behaviors that may put the participant at increased risk for HIV acquisition.
* Any preexisting physical or mental condition which may interfere with the participant's ability to comply with the dosing schedule and/or protocol evaluations or which may compromise the safety of the participant.
* Past or intended use over-the-counter or prescription medication (including herbal medications) within 7 days prior to dosing
* Exposure to more than 4 new investigational products within 12 months prior to the first dosing day.
* Current enrollment or recent past participation in another investigational study.
* Positive HIV antibody/antigen test.
* ALT more than or equal to (>=)1.5x upper limit of normal (ULN), Total bilirubin >=1.5x ULN (isolated total bilirubin more than (>)1.5xULN), and/or estimated creatinine clearance (eGFR) of less than (<)60 millilitre per minute (mL/min)/1.73 square meter (m^2).
* Regular use of tobacco or nicotine-containing products, regular alcohol consumption and/or use of known drugs of abuse.
* QT interval corrected for heart rate according to Fridericia's formula (QTcF) >450 msec.
* Evidence of previous myocardial infarction, any conduction abnormality, any significant arrhythmia, non-sustained or sustained ventricular tachycardia, and/or sinus pauses (>3 seconds).
* The participant has a tattoo or other dermatological condition overlying the location of injection or a prior history of silicone implants or fillers which may interfere with interpretation of ISRs or administration of study product.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 168 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2028-08-16 (Estimated); Study Completion 2028-08-16 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs), including Injection Site Reaction (ISR) AEs, as per severity of Grade 2-5 using the DAIDS grading scale | Up to Week 78
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. Severity of AEs and ISR AEs including injection site pain (or tenderness), erythema (or redness), induration (or swelling), and pruritis, will be assessed using Division of Acquired Immunodeficiency Syndrome (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, where Grade 1=mild, Grade 2=moderate, Grade 3=severe, Grade 4=potentially life threatening and Grade 5=Death.
Area under the plasma-concentration time curve from time zero to infinity (AUC0-inf) of VH4011499 for SAD group | Up to Week 78
Area under the plasma concentration vs time curve (AUC0-tau) for MAD group | Up to Week 78
Maximum observed plasma concentration (Cmax) of VH4011499 | Up to Week 78
Time to maximum observed plasma concentration (tmax) of VH4011499 | Up to Week 78
Apparent terminal half-life (t1/2) of VH4011499 | Up to Week 78

SECONDARY OUTCOMES:
Absolute values of liver chemistry parameters: total bilirubin and direct bilirubin (micromoles per liter [umol/L]) for SAD group | At Day 4, Day 10, Week 4, Week 24 and Week 48
Absolute values of liver chemistry parameters: total bilirubin and direct bilirubin (micromoles per liter [umol/L]) for MAD group | At Day 4, Day 10, Day 29, Day 32, Day 38, Week 24 and Week 52
Change from baseline in liver chemistry parameters: total bilirubin and direct bilirubin (umol/L) for SAD group | At Day 4, Day 10, Week 4, Week 24 and Week 48 compared to Baseline (Prior to Day 1)
Change from baseline in liver chemistry parameters: total bilirubin and direct bilirubin (umol/L) for MAD group | At Day 4, Day 10, Day 29, Day 32, Day 38, Week 24 and Week 52 compared to Baseline (Prior to Day 1)
Number of participants with maximum toxicity grade change from baseline in liver chemistry parameters: total bilirubin, direct bilirubin, alkaline phosphatase (ALP), aspartate aminotransferase (AST), and alanine aminotransferase (ALT) | Baseline (Prior to Day 1) and Up to Week 78
Absolute values of liver chemistry parameters: ALP, AST, and ALT (International Units per Liter [IU/L]) for SAD group | At Day 4, Day 10, Week 4, Week 24 and Week 48
Absolute values of liver chemistry parameters: ALP, AST, and ALT (International Units per Liter [IU/L]) for MAD group | At Day 4, Day 10, Day 29, Day 32, Day 38, Week 24 and Week 52
Change from Baseline in Liver Chemistry Parameters: ALP, AST, and ALT (IU/L) for SAD group | At Day 4, Day 10, Week 4, Week 24 and Week 48 compared to Baseline (Prior to Day 1)
Change from Baseline in Liver Chemistry Parameters: ALP, AST, and ALT (IU/L) for MAD group | At Day 4, Day 10, Day 29, Day 32, Day 38, Week 24 and Week 52 compared to Baseline (Prior to Day 1)
Number of participants with Grade 1 AEs (including ISR AEs) as per severity using the DAIDS grading scale | Week 78 post dose (Week 82 for MAD Group)
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. Severity of AEs and ISR AEs including injection site pain (or tenderness), erythema (or redness), induration (or swelling), and pruritis, will be assessed using Division of Acquired Immunodeficiency Syndrome (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, where Grade 1=mild, Grade 2=moderate, Grade 3=severe, Grade 4=potentially life threatening and Grade 5=Death.
Duration of ISR (Days) AEs by grade using the DAIDS grading scale | Week 78 post dose (Week 82 for MAD Group)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Austin, Texas

IPD SHARING:
Plan to Share IPD: Yes
Study Sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.viiv-studyregister.com/documents/About_ViiV_Patient_Level_Data_Sharing_Final_25Sep2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.viiv-studyregister.com/documents/About_ViiV_Patient_Level_Data_Sharing_Final_25Sep2023.pdf